CLINICAL TRIAL: NCT02453048
Title: Phase Ib (High Dose), Single Centre, Dose-escalating, Placebo-controlled, Randomized Study of a Live Attenuated B. Pertussis Strain Given as a Single Intranasal Dose to Healthy Adult Volunteers
Brief Title: Study of BPZE1 (High Dose) Nasal Live Attenuated B. Pertussis Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C14-80; 2015-001287-20 (EudraCT Number)
Record Dates: First submitted 2015-05-18; First posted 2015-05-25 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2018-01

CONDITIONS: Pertussis; Whooping Cough
Keywords: Pertussis; Colonization; Vaccine; Immune response; BPZE1; Infection; Bordetella pertussis; B. pertussis; respiratory Tract Infection
MeSH Terms: conditions — Whooping Cough; Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BPZE1 - 10,000,000 cfu (Experimental): Individuals will be vaccinated once intranasally with the designated dose of BPZE1 or Placebo at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  Interventions: Biological: BPZE1; Other: Placebo
- BPZE1 - 100,000,000 cfu (Experimental): Individuals will be vaccinated once intranasally with the designated dose of BPZE1 or Placebo at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  Interventions: Biological: BPZE1; Other: Placebo
- BPZE1 - 1,000,000,000 cfu (Experimental): Individuals will be vaccinated once intranasally with the designated dose of BPZE1 or Placebo at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  Interventions: Biological: BPZE1; Other: Placebo
- BPZE1 - High Antibody 1,000,000,000 cfu (Experimental): Individuals will be vaccinated once intranasally with the designated dose of BPZE1 at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  Interventions: Biological: BPZE1

INTERVENTIONS:
Biological: BPZE1 — Intranasal live, attenuated vaccine
Other: Placebo — Diluent
  Arms: BPZE1 - 1,000,000,000 cfu; BPZE1 - 10,000,000 cfu; BPZE1 - 100,000,000 cfu

SUMMARY:
This study evaluates the safety and immunogenicity of a higher dose formulation of a new live attenuated vaccine, BPZE1, intended to prevent Bordetella pertussis nasopharyngeal colonization and pertussis disease, and investigates whether higher doses of BPZE1 induce the live vaccine to colonize subjects' nasopharynx. The study is a Phase Ib (high dose), single centre, dose-escalating, placebo-controlled study of the live attenuated B. pertussis strain BPZE1 given as a single intranasal dose to healthy adult volunteer.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individual between 18 and 32 years of age, vaccinated or unvaccinated with acellular pertussis vaccine.
2. Female subject of child bearing potential must be willing to ensure that they use a highly efficient method of contraception during the study (e.g. contraceptive pill, intrauterine contraceptive device).
3. Informed consent form (ICF) signed by the subject.
4. Subject shall be able to attend all scheduled visits and to understand and comply with the study procedures.

Exclusion Criteria:

1. Individual with PT and/or PRN serum IgG antibodies ≥20 International units/ml (IU/ml). NOTE! One control group with PRN serum IgG antibodies ≥ 20 IU/ml will be included.
2. Vaccinated with the study vaccine in the Child Innovac study (EudraCT number 2010-019936-11).
3. Pregnant or lactating women. Pregnancy not planned and to be avoided during the study by use of effective contraceptive methods.
4. Blood pressure after resting ≥ 150/90 mm Hg at screening.
5. Heart rate after resting ≥ 80 bpm at screening.
6. Respiratory rate after resting ≥ 20/minute at screening.
7. Unwillingness to refrain from the use of nicotine products from screening through day 28.
8. Use of narcotic drugs and/or a history of drug/alcohol abuse with in the past 2 years prior to screening
9. The subject has donated blood or suffered from blood loss of at least 450 ml (1 unit of blood) within 60 days prior to screening or donated plasma within 14 days prior to screening.
10. Receipt of immunoglobulin, blood derived products, systemic corticosteroids or other immunosuppressant drugs within 90 days prior to day 0.
11. Asthma or other chronic respiratory problems.
12. Use of corticosteroids in the respiratory tract (e.g. nasal steroids, inhaled steroids) with in 30 days prior to day 0.
13. Receipt of a vaccine within the last 30 days prior to day 0 or planned vaccination with in the next 30 days after day 0.
14. Known hypersensitivity to any component of the study vaccine.
15. Current participation in any other clinical trial or participation (and during the whole study) in any clinical trial in the previous 3 months prior to day 0.
16. Inability to adhere to the protocol, including plans to move from the area.
17. Family (first degree) history of congenital or hereditary immunodeficiency.
18. Past or present infection with HIV, hepatitis B or C.
19. Chronic conditions requiring ongoing active medical interventions, such as diabetes mellitus or cardiovascular disease.
20. Any autoimmune or immunodeficiency disease/condition (inherited or iatrogenic).
21. Any medical condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or might affect the safety of the individual, e.g. evolving encephalopathy not attributable to another identifiable cause within 7 days of administration of a previous dose of any vaccine, hospitalization due to major depression or history of suicidal attempt.
22. Abnormal laboratory values outside the limit of normal values for the screening laboratory with clinical significance at the discretion of the investigator.
23. Person in frequent contact with children less than 1 year of age (parent, childcare worker, nurse, etc) or residence in the same household as persons with known immunodeficiency including persons on immunosuppressant therapy.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Al-Tawil, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorstensson R, Trollfors B, Al-Tawil N, Jahnmatz M, Bergstrom J, Ljungman M, Torner A, Wehlin L, Van Broekhoven A, Bosman F, Debrie AS, Mielcarek N, Locht C. A phase I clinical study of a live attenuated Bordetella pertussis vaccine--BPZE1; a single centre, double-blind, placebo-controlled, dose-escalating study of BPZE1 given intranasally to healthy adult male volunteers. PLoS One. 2014 Jan 8;9(1):e83449. doi: 10.1371/journal.pone.0083449. eCollection 2014. PMID 24421886
- [Background] Jahnmatz M, Amu S, Ljungman M, Wehlin L, Chiodi F, Mielcarek N, Locht C, Thorstensson R. B-cell responses after intranasal vaccination with the novel attenuated Bordetella pertussis vaccine strain BPZE1 in a randomized phase I clinical trial. Vaccine. 2014 Jun 5;32(27):3350-6. doi: 10.1016/j.vaccine.2014.04.048. Epub 2014 Apr 29. PMID 24793938
- [Background] Feunou PF, Kammoun H, Debrie AS, Locht C. Heterologous prime-boost immunization with live attenuated B. pertussis BPZE1 followed by acellular pertussis vaccine in mice. Vaccine. 2014 Jul 23;32(34):4281-8. doi: 10.1016/j.vaccine.2014.06.019. Epub 2014 Jun 17. PMID 24950361
- [Background] Kammoun H, Feunou PF, Foligne B, Debrie AS, Raze D, Mielcarek N, Locht C. Dual mechanism of protection by live attenuated Bordetella pertussis BPZE1 against Bordetella bronchiseptica in mice. Vaccine. 2012 Aug 31;30(40):5864-70. doi: 10.1016/j.vaccine.2012.07.005. Epub 2012 Jul 17. PMID 22814407
- [Background] Fedele G, Bianco M, Debrie AS, Locht C, Ausiello CM. Attenuated Bordetella pertussis vaccine candidate BPZE1 promotes human dendritic cell CCL21-induced migration and drives a Th1/Th17 response. J Immunol. 2011 May 1;186(9):5388-96. doi: 10.4049/jimmunol.1003765. Epub 2011 Mar 23. PMID 21430219
- [Background] Skerry CM, Mahon BP. A live, attenuated Bordetella pertussis vaccine provides long-term protection against virulent challenge in a murine model. Clin Vaccine Immunol. 2011 Feb;18(2):187-93. doi: 10.1128/CVI.00371-10. Epub 2010 Dec 8. PMID 21147936
- [Background] Feunou PF, Kammoun H, Debrie AS, Mielcarek N, Locht C. Long-term immunity against pertussis induced by a single nasal administration of live attenuated B. pertussis BPZE1. Vaccine. 2010 Oct 8;28(43):7047-53. doi: 10.1016/j.vaccine.2010.08.017. Epub 2010 Aug 13. PMID 20708998
- [Background] Feunou PF, Bertout J, Locht C. T- and B-cell-mediated protection induced by novel, live attenuated pertussis vaccine in mice. Cross protection against parapertussis. PLoS One. 2010 Apr 15;5(4):e10178. doi: 10.1371/journal.pone.0010178. PMID 20419113
- [Background] Mielcarek N, Debrie AS, Mahieux S, Locht C. Dose response of attenuated Bordetella pertussis BPZE1-induced protection in mice. Clin Vaccine Immunol. 2010 Mar;17(3):317-24. doi: 10.1128/CVI.00322-09. Epub 2010 Jan 27. PMID 20107007
- [Background] Skerry CM, Cassidy JP, English K, Feunou-Feunou P, Locht C, Mahon BP. A live attenuated Bordetella pertussis candidate vaccine does not cause disseminating infection in gamma interferon receptor knockout mice. Clin Vaccine Immunol. 2009 Sep;16(9):1344-51. doi: 10.1128/CVI.00082-09. Epub 2009 Jul 22. PMID 19625486
- [Background] Feunou PF, Ismaili J, Debrie AS, Huot L, Hot D, Raze D, Lemoine Y, Locht C. Genetic stability of the live attenuated Bordetella pertussis vaccine candidate BPZE1. Vaccine. 2008 Oct 23;26(45):5722-7. doi: 10.1016/j.vaccine.2008.08.018. Epub 2008 Aug 30. PMID 18762220
- [Derived] Jahnmatz M, Richert L, Al-Tawil N, Storsaeter J, Colin C, Bauduin C, Thalen M, Solovay K, Rubin K, Mielcarek N, Thorstensson R, Locht C; BPZE1 study team. Safety and immunogenicity of the live attenuated intranasal pertussis vaccine BPZE1: a phase 1b, double-blind, randomised, placebo-controlled dose-escalation study. Lancet Infect Dis. 2020 Nov;20(11):1290-1301. doi: 10.1016/S1473-3099(20)30274-7. Epub 2020 Jul 17. PMID 32687804
- [Derived] Lin A, Apostolovic D, Jahnmatz M, Liang F, Ols S, Tecleab T, Wu C, van Hage M, Solovay K, Rubin K, Locht C, Thorstensson R, Thalen M, Lore K. Live attenuated pertussis vaccine BPZE1 induces a broad antibody response in humans. J Clin Invest. 2020 May 1;130(5):2332-2346. doi: 10.1172/JCI135020. PMID 31945015

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Individuals will be vaccinated once intranasally with the designated dose of Placebo at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  Placebo: Diluent
- BPZE1 - 10,000,000 Cfu; BPZE1 - 100,000,000 Cfu; BPZE1 - 1,000,000,000 Cfu: Individuals will be vaccinated once intranasally with the designated dose of BPZE1 at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  BPZE1: Intranasal live, attenuated vaccine
- BPZE1 - High Antibody 1,000,000,000 Cfu: Individuals with high baseline antibodies will be vaccinated once intranasally with the designated dose of BPZE1 at a Dose 2 x 0.4 mL (0.4 mL per nostril).
  BPZE1: Intranasal live, attenuated vaccine
Period: Overall Study
Arm/Group | Placebo | BPZE1 - 10,000,000 Cfu | BPZE1 - 100,000,000 Cfu | BPZE1 - 1,000,000,000 Cfu | BPZE1 - High Antibody 1,000,000,000 Cfu
Started | 12 | 12 | 12 | 12 | 6
6-month Follow-up | 12 | 12 | 12 | 12 | 6
Completed | 12 | 11 | 10 | 12 | 0
Not Completed | 0 | 1 | 2 | 0 | 6
Not completed — Only part of initial 6 mo. study | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BPZE1 - 10,000,000 Cfu | BPZE1 - 100,000,000 Cfu | BPZE1 - 1,000,000,000 Cfu | BPZE1 - High Antibody 1,000,000,000 Cfu | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 6 | 54
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 2 | 0 | 0 | 0 | 0 | 2
  20-25 years | 3 | 2 | 4 | 3 | 2 | 14
  25-30 years | 7 | 7 | 7 | 6 | 4 | 31
  >=30 years | 0 | 3 | 1 | 3 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 2 | 7 | 1 | 21
  Male | 6 | 7 | 10 | 5 | 5 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 12 | 6 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 12 | 12 | 12 | 12 | 6 | 54
Height [Median (Inter-Quartile Range); unit: m] | 1.74 [1.63 to 1.85] | 1.77 [1.72 to 1.88] | 1.8 [1.75 to 1.83] | 1.72 [1.67 to 1.77] | 1.76 [1.72 to 1.8] | 1.76 [1.72 to 1.80]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 22 [20 to 24] | 22 [22 to 25] | 22 [20 to 28] | 23 [22 to 26] | 22 [20 to 24] | 22 [21 to 25]
Weight [Median (Inter-Quartile Range); unit: kg] | 69 [59 to 77] | 71 [64 to 84] | 74 [63 to 93] | 69 [61 to 81] | 69 [60 to 79] | 70 [62 to 82]
Oral Temperature [Median (Inter-Quartile Range); unit: C] | 36.5 [36.4 to 36.9] | 36.8 [36.6 to 37.0] | 36.6 [36.3 to 36.9] | 36.6 [36.2 to 37.0] | 36.3 [35.9 to 36.5] | 36.6 [36.4 to 36.9]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint is the Number and Percentage of Participants Per Dose Group and Randomized Allocation, With at Least One of the Following Adverse Events Between Day 0 and Day 28
Description: Percentage is based on subjects experiencing at least one of the following events:
  * Cough and spasmodic cough of grade 2 or higher
  * Other respiratory tract AE related or possibly related to vaccination of grade 3 or higher
  * Any other AE related or possibly related to vaccination of grade 3 or higher
Time Frame: 28 days
Population: Arms (Placebo separated from randomized groups)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Subjects receiving intranasal Placebo
- Low Dose Group: Subjects receiving 10^7 CFU of intranasal BPZE1
- Medium Dose Group: Subjects receiving 10^8 CFU of intranasal BPZE1
- High Dose Group: Subjects receiving 10^9 CFU of intranasal BPZE1
- PRN High Group: Subjects with a pre-existing baseline PRN > 20 IU that received 10^9 CFU of intranasal BPZE1 (non-randomized group)
Arm/Group | Placebo | Low Dose Group | Medium Dose Group | High Dose Group | PRN High Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 6
Participants
  Cough or Spasmodic Cough of grade >=2 | 1 | 1 | 1 | 2 | 0
  Other respiratory tract AE of grade >=3 | 0 | 0 | 1 | 1 | 0
  Other AE grade >=3 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Subjects With BPZE1 Colonization
Description: To assess the proportion of subjects having positive colonization of the human respiratory tract by live attenuated B. pertussis strain BPZE1 per group at any time period measured at 4, 7, 11, 14, 21 and 28 days post vaccination.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose Group | Medium Dose Group | High Dose Group | PRN High Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 6
Participants
  Colonized | 0 | 10 | 9 | 10 | 2
  Not Colonized | 12 | 2 | 3 | 2 | 4

3. Secondary Outcome: The Proportion of Subjects That Have an Antibody Response to BPZE1 Vaccination
Description: To assess the number of immune responders and levels of Immunoglobulin G/Immunoglobulin A (IgG/IgA) antibodies to pertussis toxin (PT), filamentous haemagglutinin adhesin (FHA), Pertactin (PRN), and fimbriae 2/3 in serum and nasopharyngeal aspirate.
  A positive antibody response after vaccination is defined as at least 100% increase from pre- to post-vaccination, to at least 4 times minimum level of detection (MLD) for PT, FHA, PRN, and fimbriae 2/3 in the post-vaccination sample. The 4 antigens described are the standard 4 antigens historically used to describe a serum immunological response to B. pertussis. The absolute serum antibody titers have not shown a correlation of protection in previous pertussis vaccine studies of the current acellular vaccine and there is no known serum antigen threshold of protection for pertussis.
  Antibodies are measured before vaccination and at 4, 7, 11, 14, 21, 28 days, 6-months and 12-months post-vaccination.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose Group | Medium Dose Group | High Dose Group | PRN High Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 6
Participants
  IgG Response: Non-responding Subjects | 11 | 1 | 4 | 1 | 2
  IgG Response: 1 Antigen | 1 | 3 | 2 | 4 | 1
  IgG Response: 2 Antigens | 0 | 1 | 2 | 3 | 2
  IgG Response: 3 Antigens | 0 | 4 | 2 | 3 | 1
  IgG Response: 4 Antigens | 0 | 3 | 2 | 1 | 0
  IgA Response: Non-responding Subjects | 10 | 3 | 5 | 2 | 2
  IgA Response: 1 Antigen | 2 | 1 | 2 | 1 | 1
  IgA Response: 2 Antigens | 0 | 3 | 1 | 6 | 2
  IgA Response: 3 Antigens | 0 | 3 | 4 | 3 | 1
  IgA Response: 4 Antigens | 0 | 2 | 0 | 0 | 0
  IgG or IgA Response: Non-responding Subjects | 10 | 1 | 3 | 0 | 2
  IgG or IgA Response: 1 Antigen | 2 | 3 | 2 | 1 | 0
  IgG or IgA Response: 2 Antigens | 0 | 1 | 0 | 4 | 1
  IgG or IgA Response: 3 Antigens | 0 | 4 | 4 | 4 | 2
  IgG or IgA Response: 4 Antigens | 0 | 3 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: 14 days, 1 month, 3 months, 6 months, 1 year
Arm/Group | Placebo | Low Dose Group | Medium Dose Group | High Dose Group | PRN High Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 1/12 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12 | 11/12 | 9/12 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Low Dose Group (N=12) | Medium Dose Group (N=12) | High Dose Group (N=12) | PRN High Group (N=6)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Low Dose Group (N=12) | Medium Dose Group (N=12) | High Dose Group (N=12) | PRN High Group (N=6)
Cough - week 1 (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 2 | 1
Cough - week 2 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 0
Fatigue - week 1 (General disorders) | 6 | 5 | 6 | 4 | 4
Fatigue - Week 2 (General disorders) | 1 | 2 | 2 | 1 | 1
Headache - week 1 (Nervous system disorders) | 5 | 2 | 6 | 3 | 3
Headache - week 2 (Nervous system disorders) | 0 | 2 | 1 | 3 | 0
Nasal Congestion - week 1 (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 4 | 2 | 3
Nasal Congestion - week 2 (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 0 | 1
Rhinorrhoea - week 1 (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4 | 3 | 2
Rhinorrhoea - week 2 (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1 | 0
Sneezing - week 1 (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 4 | 6 | 2
Sneezing - week 2 (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications will be co-authored by the PI and the Sponsor (Inserm).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT02453048/Prot_SAP_000.pdf